CLINICAL TRIAL: NCT04395014
Title: Echocardiographic Assessment of Ventricular Strain During a Healthy Pregnancy in the First, Second, and Third Trimester.
Acronym: VStrain123P
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Miguel Ayala León (Network)
Collaborators: Leiden University Medical Center (Other); Institute of Security and Social Services of Workers of the State of Puebla. (Unknown)
Responsible Party: Sponsor-Investigator, Miguel Ayala León, cardiovascular critical care unit director, Hospital Beneficencia Espanola de Puebla
Organization: Hospital Beneficencia Espanola de Puebla (Network)
Other Study IDs: Cardiology-003
Record Dates: First submitted 2020-05-14; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Echocardiography; Pregnancy Related Conditions, Unspecified, First Trimester; Pregnancy Related Conditions, Unspecified, Second Trimester; Pregnancy Related Conditions, Unspecified, Third Trimester; Ventricle Remodeling
Keywords: Strain ventricular; Pregnancy; Ventricular function
MeSH Terms: conditions — Ventricular Remodeling | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2D Echocardiography — In this echocardiographic imaging acquisition protocol, the pregnancy patients, are colocated in the left lateral decubitus position on a clinical bed with the left arm flex and the hand behind the head. All the echocardiographic measurements are taken by the examiner in this position.

SUMMARY:
Pregnancy is a physiological situation that produces transient preload and afterload changes. The heart is subjected to reversible morphological remodelings and hemodynamic and functional adaptations. The characterization and understanding of maternal cardiac function during normal pregnancy by echocardiography 2D is of clinical importance for the opportune recognition of cardiac pathology.

This study aims to investigate pregnancy-induced changes in ventricular strain in healthy pregnant women by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and < 35
* Patients who coursing the first trimester of pregnancy
* No history or symptoms of cardiovascular or lung disease
* No ongoing or previous cardio or vasoactive treatment
* Normal ECG
* Normal physical examination
* Able to give informed consent

Exclusion Criteria:

* Poor acoustic window
* Obesity in the first trimester (body mass index [BMI], ≥30 kg/m2)
* Inability to provide consent.
* Tricuspid regurgitation more than mild
* Collagen disease
* Professional sports activity
* Twin pregnancy
* Hyperthyroidism

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women that coursing the first trimester of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular telediastolic diameter (LVTDd) | 3 minutes
  Left ventricular telediastolic diameter (mm)
Left ventricular telesystolic diamete (LVTSd) | 3 minutes
  Left ventricular telesystolic diameter (mm)
Interventricular septum (IVS) | 3 minutes
  Diameter of Interventricular septum (mm)
Left ventricular posterior wall (LVPW) | 3 minutes
  Left ventricle posterior wall (mm)
Ejection fraction (EF) | 3 minutes
  Ejection fraction (%)
Right atrium area (RA area) | 3 minutes
  Right atrium area (cm2)
Right ventricle B | 3 minutes
  Right ventricle basal dimension (mm)
Right ventricular M | 3 minutes
  Right ventricle mid cavity dimension (mm)
Right ventricular L | 3 minutes
  Right ventricle longitudinal dimension (mm)
Right ventricle outflow tract dimension at the proximal subvalvular level (RVOT p) | 3 minutes
  Right ventricle outflow tract dimension at the proximal subvalvular level (mm)
Right ventricle outflow tract dimension at the distal or pulmonic valve level (RVOT d) | 3 minutes
  Right ventricle outflow tract dimension at the distal or pulmonic valve level (mm)
Tricuspid annular plane systolic excursion (TAPSE) | 3 minutes
  Tricuspid annular plane systolic excursion (mm)
Right ventricle free wall (RV free wall) | 3 minutes
  Right ventricle free wall (mm)
Inferior cava vein (ICV) | 3 minutes
  Inferior cava vein (mm)
Left atrium volume index (LA volume index) | 3 minutes
  Left atrium volume index (mL/m2)
E mitr | 3 minutes
  Mitral E wave (cm/s)
A mitr | 3 minutes
  Mitral A wave (cm/s)
E/A mitr | 3 minutes
  Mitral E wave / Mitral A wave
Sm | 3 minutes
  S-wave at mitral anulus (cm/s)
Em | 3 minutes
  E-wave at mitral annulus (cm/s)
Am | 3 minutes
  A-wave at mitral annulus (cm/s)
Em/Am | 3 minutes
  E-wave at mitral annulus/ A-wave at mitral annulus
E/Em | 3 minutes
  E wave/ E-wave at the mitral annulus
E tric | 3 minutes
  Tricuspid E wave (cm/s)
A tric (cm/s) | 3 minutes
  Tricuspid A wave (cm/s)
E/A tric | 3 minutes
  Tricuspid E wave/Tricuspid A wave
St | 3 minutes
  S-wave at tricuspid anulus(cm/s)
Et | 3 minutes
  E-wave at tricuspid anulus(cm/s)
At | 3 minutes
  A-wave at tricuspid anulus (cm/s)
Et/At | 3 minutes
  E-wave at tricuspid anulus /A-wave at tricuspid anulus
Mean pulmonary artery pressure (mPAP) | 3 minutes
  Mean pulmonary artery pressure (mmHg)
Systolic pulmonary artery pressure (sPAP) | 3 minutes
  Systolic pulmonary artery pressure (mmHg)
Stroke volume (SV) | 3 minutes
  Stroke volume (mL)
Cardiac output (CO) | 3 minutes
  Cardiac output (L/min)
Strain right ventricle (Strain RV) | 3 minutes
  Strain right ventricle
Strain left ventricle (Strain LV) | 3 minutes
  Strain left ventricle

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beneficencia Española de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No